CLINICAL TRIAL: NCT00728442
Title: Impact of the OncoDoc2 Decision Support System on Compliance of Multidisciplinary Staff Meeting Decisions With Clinical Practice Guidelines in the Management of Non-metastatic Breast Cancer.
Brief Title: Impact of OncoDoc2 on Guideline Compliance in the Management of Breast Cancer
Acronym: OncoDoc2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: K 070603
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Clinical practice guidelines; Guideline adherence; Clinical decision support systems; Randomized controlled trial; Intervention study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): medical decision based on computerized guideline-based decision support system
  Interventions: Device: ONCODOC LOGICIEL
- 2 (No Intervention)

INTERVENTIONS:
Device: ONCODOC LOGICIEL — Introduction of a computer-based decision support system in the medical decision process
  Arms: 1

SUMMARY:
The objective of the study is to evaluate how the use of OncoDoc2, a computerized guideline-based decision support system, could improve the compliance of multidisciplinary staff meeting decisions with local clinical practice guidelines in the management of non-metastatic breast cancer.

DETAILED DESCRIPTION:
In France, to promote the quality of cancer care, decisions have currently to be made according to clinical practice guidelines (CPGs) during regularly organized multidisciplinary staff meetings (MSMs). Dissemination of textual CPGs has a poor impact on clinical practice as opposed to the use of clinical decision support systems (CDSSs) known to improve compliance with CPGs. OncoDoc2 is a CDSS providing patient-specific recommendations based on CPGs for non-metastatic female breast cancer management elaborated by the CancerEst INTERMEDICAL collaboration.The main goal of the study is to evaluate the effect of the routine use of OncoDoc2 during MSMs on compliance of MSM decisions with local CPGs. Impact will be measured by the compliance rate of MSM decisions with OncoDoc2 recommendations. The design of the study relies on a cluster randomized controlled trial. Under the assumption of a baseline compliance rate of 70% without intervention, an expected compliance rate of 90% in the intervention group (α = 5%, β = 20%), an inter-cluster variability of 5%, and 59 decisions per center, the required number of centers is 3 in each group, or 177 decisions in each arm. The study will be conducted in cancer care centers (public and private) from Paris area, France.This prospective trial will be conducted in two steps. First, baseline compliance rates will be measured in each center. Then, the 6 centers will be randomized into 2 arms. In the intervention arm, OncoDoc2 will be used during MSMs at decision time. Every case of non-adherence with system recommendations will have to be justified by clinicians. In both arms and after each MSM, MSM decisions will be recorded as well as patient characteristics and OncoDoc2 will be used for each patient case to get system recommendations. In the intervention arm, OncoDoc2 recommendations obtained by MSM will also be recorded, as well as the reason for non following recommendations in case MSM decision does not comply with guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Non metastatic, including invasive and in situ, breast cancers as well as axillary cancer without breast tumor.
* At least one therapeutic MSM decision.

Exclusion Criteria:

* Breast disease without cancer
* Metastatic breast cancer
* Male breast cancer
* Breast cancer cases when medical records are not accessible to investigators
* Management but not therapeutic breast cancer decisions (diagnostic investigations, treatment follow-up, delayed decisions…)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Compliance of multidisciplinary staff meeting (MSM) decisions with OncoDoc2 guideline-based recommendations at one year : MSM decisions are recorded on a weekly basis. | Every week

SECONDARY OUTCOMES:
Compliance of actually administered treatments with OncoDoc2 recommendations at 18 months (treatments administration may last until 8 months after the therapeutic decision has been taken by MSMs) | at 18 months
typology of non-compliant reasons for both MSM decisions and treatments administration | at 18 months
patient profiles associated with non-guideline-compliant therapeutic decisions. | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge UZAN, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de gynecologie obstetrique, Hopital Tenon, Paris, France